CLINICAL TRIAL: NCT06542471
Title: Dual Intramedullary Nailing Fixation Versus Dual Plating of Pediatric Both Bone Forearm Fracture: a Study Protocol for a Randomized Controlled Trial
Brief Title: Plating Versus Nailing in Pediatric BB Forearm Fractures
Acronym: DINDPL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23ew234
Record Dates: First submitted 2024-07-06; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Intramedullary Nail; Plate Fixation; Forearm Fracture; Randomized Controlled Trial
Keywords: forearm fractures; pediatric fractures; flexible nail; plate fixation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Intramedullary nail group
  Interventions: Device: Dual intramedullary nailing
- group 2 (Experimental): Plating group
  Interventions: Device: Dual plating

INTERVENTIONS:
Device: Dual intramedullary nailing — - Elastic nailing for radius under image guidance through distal entry point and physeal sparing technique.
  Arms: group 1
Device: Dual plating — - ORIF for radius done first through volar approach.
  Arms: group 2

SUMMARY:
A randomized controlled trial to compare between dual intramedullary nailing and dual plating trying to synthesis a high quality evidence study that can solve the conflict between the decisions.

ELIGIBILITY:
Inclusion criteria:

1. Both-bone Forearm Diaphyseal Fracture.
2. age more than or equal nine years old with open distal radius physis.
3. Simple transverse or short oblique fractures (2R2-A2,2R2-A3,2U2-A2,2U2-A3) according to OTA/ AO classification.

Exclusion criteria:

1. Neurovascular injury.
2. Open fractures
3. Comminuted fractures
4. Pathological fractures

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to union | 6 months
  weeks required to achieve union
Elbow range of motion | 6 months
  elbow flexion, extension, pronation and supination in degrees
Quick DASH score | 6 months
  Patient reported questionnaire
patient satisfaction questionnaire | 6 months
  five points Likert scale

SECONDARY OUTCOMES:
Adverse events | 6 months
  Any adverse event will be recorded
Re-operation rate | 6 months
  percentage of patients requiring reoperation
size of wound scar in millimeters | 6 months
  measuring the size of wound scar in millimeters
Deformity (malunion rate) | 6 months
  Malunion deformity

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Mahran, MD, Study Chair — Ain Shams University; Ahmed Saeed Younis, Study Director — Ain Shams University; Abdelrahman Hani, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt